CLINICAL TRIAL: NCT01040741
Title: A Prospective Observational Study of Safety and Occurrence of Influenza-like Illness Following Administration of Adjuvanted Swine Origin A(H1N1) Pandemic Subunit Vaccine Focetria
Brief Title: Observational Safety Study of Adjuvanted Swine Origin A (H1N1) Pandemic Subunit Egg Derived Vaccine
Status: Completed | Type: Observational
Sponsor: Novartis Vaccines (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Other Study IDs: V111_09OB
Record Dates: First submitted 2009-12-29; First posted 2009-12-30 (Estimated); Last update posted 2011-10-05 (Estimated); Status verified 2011-10

CONDITIONS: Pandemic Influenza A (H1N1); A New Flu Virus of Swine Origin
Keywords: Pandemic influenza A (H1N1) vaccine; Adjuvanted

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (6):
- Group 1: 6-23 months
  Interventions: Other: Non-intervention observational study
- Group 2: 2-8 years
  Interventions: Other: Non-intervention observational study
- Group 3: 9-17 years
  Interventions: Other: Non-intervention observational study
- Group 4: 18-44 years
  Interventions: Other: Non-intervention observational study
- Group 5: 45-60 years
  Interventions: Other: Non-intervention observational study
- Group: >60 years
  Interventions: Other: Non-intervention observational study

INTERVENTIONS:
Other: Non-intervention observational study — Non-intervention observational study

SUMMARY:
This is an observational safety study of a prophylactic use of Flu Egg Derived Adjuvanted Swine Origin A(H1N1) Vaccine in subjects 6 months of age and older. Subjects may receive either 1 or 2 doses: children and elderly will receive 2 doses and adults will receive either 1 or 2 doses.

ELIGIBILITY:
Inclusion Criteria:

* Subject's age in accordance with the approved product label of the country where the study is conducted
* Subjects will be vaccinated with Focetria®, independently of this study.
* Subjects or parent/guardian willing to provide informed consent prior to vaccination administration and complete all of the study, including follow-up contact

Exclusion Criteria:

• Received any prior H1N1 vaccination

Min Age: 6 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Population of children, adolescents, adults and elderly
Sampling Method: Non-Probability Sample
Enrollment: 7284 (Actual)
Dates: Start 2009-12; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
To quantify the safety of Flu Egg Derived Adjuvanted Swine Origin A(H1N1) Pandemic Subunit Vaccine in actively monitored subjects; To characterize the incidence of AEs in specific age groups following an active surveillance of vaccinated subjects. | 6 Months

SECONDARY OUTCOMES:
To assess the occurrence of laboratory confirmed H1N1sw and influenza-like illness following vaccination with Flu Egg Derived Adjuvanted Swine Origin A(H1N1) Pandemic Subunit Vaccine. | 6 months

CONTACTS AND LOCATIONS:
Locations (14):
- Argentina (6):
  - Hospital Garrahan, Combate de Los Pozos 1881, Buenos Aires F.D.
  - Hospital de Ninos "Dr. Ricardo Gutierrez", Gallo 1330, Buenos Aires F.D.
  - Hospital Nuestra Señora de la Misericordia, Belgrano 1500, Córdoba Province
  - Hospital Pediatrico del Niño Jesus, Castro Barros 650 - San Martín, Córdoba Province
  - Sanatorio Mayo Privado S.A., Humberto Primo 520, Córdoba Province
  - Hospital Pediatrico "Dr. Humberto Notti", Bandera de Los Andes 2603 Villa Nueva, Guaymallen Mendoza
- Netherlands (8):
  - Huisartsenpraktijk Bergentheim, Kanaalweg West 61, Bergentheim
  - Huisartsenpraktijk Bredero, Brederostraat 2/A, Breda
  - Saxenburg Groep, Zorgcentrum Aleida Kramer, M.v.d. Thijnensingel 1, Coevorden
  - Huisartsenpraktijk Dennenlaan, Dennenlaan 56, Emmen
  - Huisartsenpraktijk de Steenpoort, Prinses Julianastraat 25, Genemuiden
  - Huisartsenpraktijk Gramsbergen, Voorstraat 3, Gramsbergen
  - Huisartsenpraktijk Oosterhesselen, Edveensweg 13, Oosterhesselen
  - Isala Klinieken Zwolle, Groot Wezenland 20, Zwolle